CLINICAL TRIAL: NCT01060033
Title: A Study of Novel Magnetic Resonance Imaging Sequences for Target Delineation and Prognostication in Cervical Cancer
Brief Title: MRI (Including Spectroscopy and Fat-Saturations and Diffusion-Weighted Imaging) in Cervical Cancer
Acronym: MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 10-0033 / 201109278
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Squamous cell cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Magnetic Resonance Spectroscopy; Diffusion Magnetic Resonance Imaging; Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): * Clinical T1/T2-weighted MRI sequence per standard of care before treatment, during treatment per standard protocol, and at 3 months.
  * Patients may have one or all of the following sequences in addition to the standard MRI imaging:
    * MR Spectroscopy
    * Fat-saturation and Diffusion-Weighted Imaging
    * Dynamic Contrast Enhancement MRI (MR-DCE)
    * Diffusion Tensor Imaging (DTI)
  Interventions: Device: MR Spectroscopy; Device: Fat-Saturation and Diffusion-Weighted Imaging; Device: Dynamic Contrast Enhancement MRI (MR-DCE); Device: Diffusion Tensor Imaging (DTI)

INTERVENTIONS:
Device: MR Spectroscopy
Device: Fat-Saturation and Diffusion-Weighted Imaging
Device: Dynamic Contrast Enhancement MRI (MR-DCE)
Device: Diffusion Tensor Imaging (DTI)

SUMMARY:
To detect differences in MR spectroscopy, diffusion weighted MR, diffusion tensor imaging (DTI) or dynamic contrast enhancement (DCE) MR imaging between primary cervical tumors and normal cervical tissue.

DETAILED DESCRIPTION:
At our institution, all patients receiving external beam and/or brachytherapy as part of the treatment of primary cervical cancer receive CT, PET, and MRI simulation scans as standard of care. Brachytherapy patients also receive weekly T1/T2 weighted MR simulation scans as part of their treatment planning.

We propose the use of additional MR sequences to the standard T1/T2 weighted MR simulation scans. The data obtained from these additional sequences will be used for improving tumor delineation and obtaining prognostic information.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-proven newly diagnosed squamous cell cervical cancer (FIGO clinical stages IB2-IVA).
* Patients must be ≥ 18 years of age.
* Patients must be able to receive standard radiation therapy (external beam radiation and brachytherapy) with or without chemotherapy.
* Patients with distant metastatic disease are eligible provided the estimated survival of the patient is at least one year.
* Patients must be scheduled to undergo or have already undergone FDG-PET/CT imaging for clinical staging cervical cancer at Barnes-Jewish Hospital Clinical PET facility on the Siemens Biograph 40 True Point Tomograph Scanner or elsewhere in the WUSM Nuclear Medicine department using the quality controls instituted by Nuclear Medicine.
* Patients must be able to give informed consent.

Exclusion Criteria:

* Patients with another known active malignancy.
* Patients who have received treatment for any malignancy (with the exception of non-melanoma skin cancer) in the past 5 years.
* Pregnant or breastfeeding patients.
* Patients whose tumors are not FDG avid on baseline standard of care FDG-PET/CT imaging.
* Patients with contraindications to MRI scanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Differences in MR spectroscopy, diffusion weighted MR, diffusion tensor imaging (DTI) or dynamic contrast enhancement (DCE) MR imaging between primary cervical tumors and normal cervical tissue. | 3 months

SECONDARY OUTCOMES:
Determine whether MR-DCE or MR-FS or DTI can improve target delineation in primary cervical tumors. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Esthappan, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu